CLINICAL TRIAL: NCT07090148
Title: Pilot Trial of a DNA Vaccine Encoding Prostatic Acid Phosphatase (pTVG-HP) and PD-1 Blockade, With Targeted Ablation of Resistant Lesions, in Patients With Non-Castrate Recurrent Oligometastatic Prostate Cancer
Brief Title: Trial of pTVG-HP+Nivo+Targeted Ablation of Resistant Lesions in Non-Castrate RecurrentOMPC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0825; HT94252411043 (Other Grant/Funding Number: Department of Defense); A533300 (Other: UW Madison); SMPH/HUMAN ONCOLOGY/HUMAN ONCO (Other: UW Madison); UW25025 (Other: UW Madison); Protocol Version 4/15/2025 (Other: UW Madison)
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer Patients; Non-castrate Prostate Cancer; Recurrent Prostate Cancer; Oligometastatic Prostate Cancer (OMPC)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — spartalizumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with non-castrate, recurrent, oligometastatic prostate cancer (Experimental): Participants will receive a combination of vaccine and immunotherapy.
  Interventions: Biological: pTVG-HP DNA vaccine; Drug: Anti-PD-1 monoclonal antibody

INTERVENTIONS:
Biological: pTVG-HP DNA vaccine — The vaccine will be injected into the outer side of the upper area of the arm in two adjacent sites, with 0.25 mL administered at each site.
Drug: Anti-PD-1 monoclonal antibody — Nivolumab is a potent human immunoglobulin G4 (IgG4) monoclonal antibody (mAb). Participants will receive two 10mg doses.
  Other Names: Opdivo; nivolumab

SUMMARY:
The goal of this clinical trial is to learn whether an experimental vaccine called pTVG-HP ("vaccine" or "DNA vaccine"), combined with a drug called nivolumab can increase the cancer-fighting ability of a person's immune cells.

The main question it aims to answer is whether the combination of medicines can get rid of metastatic tumors in participants with non-castrate, recurrent, oligometastatic prostate cancer.

Participants will undergo:

* Treatment with pTVG-HP
* Treatment with Nivolumab
* Radiation Therapy

DETAILED DESCRIPTION:
To explore the use of an investigational DNA vaccine, pTVG-HP, a plasmid DNA encoding human prostatic acid phosphatase (PAP), in combination with nivolumab delivered with vaccination, and in combination with targeted ablation of treatment-resistant lesions, to eradicate metastatic tumor lesions in patients with non-castrate, recurrent, oligometastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age with a histologic diagnosis of adenocarcinoma of the prostate
* Participants must have undergone radical prostatectomy
* Participants must have completed local therapy by surgery, and any adjuvant/salvage radiation therapy (if required), at least 3 months prior to entry, with removal or ablation of all visible disease, including seminal vesical and/or local lymph node involvement.
* Participants must have biochemically recurrent disease defined by the following:

  * Participants must have evidence of detectable serum PSA with at least 4 serum PSA measurements available, from the same clinical laboratory, at least two weeks apart up to one year, and the final serum PSA value must be > 2.0 ng/mL.
  * PSA doubling time, calculated from most recent 4 serum PSA values (collected up to one year prior to enrollment, at least 2 weeks apart, and all from the same clinical laboratory), must be a positive number (i.e. evidence of PSA rise over time).
* Participants must have oligometastatic disease, defined as:

  * < 3 lesions consistent with metastases as detected by CT of the abdomen/pelvis and bone scintigraphy (bone scan)
  * Lesions consistent with metastatic prostate cancer as detected by PSMA PET/CT
* Participants with a prior history of a second malignancy are eligible provided they have been treated with curative intent and have been free of disease greater than three years. There will be no exclusion for patients with a history of basal cell carcinoma, squamous cell skin cancer, superficial bladder cancer, or other in situ carcinoma that has been adequately treated.
* Participants who are sexually active must use a reliable form of contraception while on study and for 4 weeks after the last immunization.
* ECOG performance score < 2 and life expectancy of at least 12 months.
* Participants must have normal hematologic, renal and liver function
* Participants must be informed of the experimental nature of the study and its potential risks and must sign an IRB-approved written informed consent form indicating such an understanding.
* Willingness to provide blood samples for immune studies, per study calendar, up to one year after study, even if off treatment.

Exclusion Criteria:

* Small cell or other variant prostate cancer histology
* Participants cannot have evidence of immunosuppression or have been treated with immunosuppressive therapy, such as chemotherapy or chronic treatment dose corticosteroids (greater than the equivalent of 10 mg prednisone per day), within 3 months of the first vaccination.
* Seropositive for HIV, hepatitis B (HBV) or hepatitis C (HCV) per patient history due to the immunosuppressive features of these diseases.
* Prior treatment with an LHRH agonist or nonsteroidal antiandrogen, except in the following circumstances: Neoadjuvant/adjuvant androgen deprivation therapy administered with radiation therapy or at the time of prostatectomy is acceptable, provided that there was no evidence of PSA progression while on treatment. In this situation, patients must not have received more than 24 months of androgen deprivation treatment. Other treatment with androgen deprivation therapy is prohibited.
* Serum testosterone at screening < 50 ng/dL.
* Participants must not be concurrently taking other medications or supplements with known hormonal effects, including PC-SPES, megestrol acetate, finasteride, ketoconazole, estradiol, or Saw Palmetto. All other medications with possible anti-cancer effects must be discussed with the PI prior to study entry.
* Participants previously treated with other potential or experimental therapies for prostate cancer must have discontinued these treatments and completed at least a 4 week washout prior to beginning treatment.
* Participants must not have known psychological or sociological conditions, addictive disorders or family problems, which would preclude compliance with the protocol.
* Participants with unstable or severe intercurrent medical conditions or laboratory abnormalities that would impart, in the judgment of the PI, excess risk associated with study participation or study agent administration.
* Participants who have concurrent enrollment on other phase I, II, or III investigational therapeutic treatment studies for prostate cancer cannot be actively receiving treatment and the last dose cannot be within 4 weeks of day 1. They must be in the follow up phase of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
PSA (prostate-specific antigen) complete response rate | 12 months
  Defined as a serum PSA <0.2 ng/mL at 1 year after prostatectomy
Incidence of Adverse Events | 5 years
  Adverse events will be evaluated using the most recent version of the Common Terminology Criteria for Adverse Events (CTCAE).
Toxicity Rates | 5 years
  Toxicity rates (grade 2, grade 3, grade 4, grade ≥ 2, grade ≥ 3, etc.) will be calculated for each study arm and reported along the corresponding 95% confidence intervals. The 95% confidence intervals will be constructed using the Wilson score method.

SECONDARY OUTCOMES:
Metastasis-free survival rate at 1 year | 12 months
Metastasis-free survival rate at 2 years | 2 years
Progression-free survival (PSA) at 5 years | 5 years
  Defined as a serum PSA <0.2 ng/mL at 5 years after prostatectomy, in patients with non-castrate (>25 ng/dL) testosterone levels.
Change in PSA doubling time | Baseline to 5 years
Change in PSA slope | Baseline to 5 years
Overall PSA response rate | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Douglas McNeel, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes